CLINICAL TRIAL: NCT01556035
Title: A Multicentre Prospective Phase II Single Arm Trial Evaluating the Benefit of Therapy With Lenalidomide (Revlimid®) in Relapsed or Refractory Primary-cutaneous Large B-cell Lymphoma (Leg-type) After First Line Treatment by Chemotherapy Plus Rituximab for the French Study Group of Cutaneous Lymphoma (GFELC)
Brief Title: Lenalidomide in Relapsed or Refractory Primary-cutaneous Large B-cell Lymphoma Leg-type : Multicentre Prospective Phase II Single Arm Trial of the French Study Group of Cutaneous Lymphoma
Acronym: REV-LEG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2011/28
Record Dates: First submitted 2012-03-12; First posted 2012-03-16 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Refractory Primary-cutaneous Large B-cell Lymphoma (Leg-type)
Keywords: oncodermatology; hematology; cutaneous B cell lymphoma; lenalidomide
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide treatment (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Patient orally treated with lenalidomide 25 mg daily for 21 days with 7 days rest of a 28 days cycle.Treatment maintained for 12 months unless progression

SUMMARY:
In spite of high initial response rate after a first line treatment by R-polychemotherapy, cutaneous but also extra-cutaneous recurrences occur after 2 years in about half of the patients with PCBCL-LT. Thereafter there is no consensus concerning patients care: radiotherapy has only a palliative effect, advanced age often limits using more aggressive chemotherapies and no treatment has demonstrated a prolonged efficacy in these relapsing cases. Therefore new alternatives therapeutic options are needed. Lenalidomide has an antineoplastic pro-apoptotic effect but also immunomodulatory, and antiangiogenic properties. Preliminary results suggest its efficacy in relapsing or refractory diffuse large B-cells lymphomas, especially of nongerminal cells phenotype. By analogy with these results, lenalidomide appears as an attractive candidate in PCLBCL-LT, more specially as it has a manageable toxicity even in advanced age patients.

If the lenalidomide efficacy is confirmed in relapsing PCLBCL-LT, this will plead its evaluation as maintenance therapy after R-chemotherapy in order to avoid recurrences.

DETAILED DESCRIPTION:
To assess benefit and safety of lenalidomide in patients with refractory or relapsing primary cutaneous large B-cell lymphoma leg type (PCBCL-LT) after a first line treatment by Rituximab and polychemotherapy. The primary endpoint is overall response rate (complete response and partial response) at 6 months. Response will be assessed according to clinical and isotopic criteria.

Optional biological study:

A biological collection (skin and blood samples) will be established. Predictive biological markers of response or of aggressiveness and resistance to the treatment will be investigated on the skin biopsies by phenotypic and genetic analyses. The recent discovery of BLIMP1 inactivation or deletion at 6q21 in activated B-cell like type of diffuse large B-cell systemic lymphoma points to the need of both a global genetic analysis by Array-CGH with Single Nucleotide Polymorphism study and a specific investigations of the status of genes such as CDKN2A, BCL2, BCL6 and BLIMP1 by FISH analysis and/or gene dosage. Xenograft will be performed from skin biopsies in order to develop animal models for PCLBCL-LT.

Lenalidomide stimulates NK cells immunity and enhances anti-tumor responses. It also seems to modify the phenotype of NK cells through a decrease of the expression of Killer cell Immunoglobulin-like Receptors and NKp46. The expression of the NK receptors on blood cells will be analyzed in order to evidence modifications of the phenotypical and functional changes under treatment, and to search for a correlation with the clinical response to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven Primary cutaneous large B-cell lymphoma leg-type
* Clinically measurable skin involvement (T1-T3) or skin and nodal (N1-N3) involvement measurable by PET-CT, corresponding to :

Relapse after initial complete response (CR) after R-polychemotherapy Or Partial response or stable disease after R-polychemotherapy

* Age > 18 years
* Life expectancy > 3 months
* WHO performance status 0-2
* Skin biopsy performed at the inclusion on a skin tumor : new tumor in case of relapsing PCLBCL-LT or initial skin tumor refractory to the previous treatment
* Signed informed consent for clinical and biological analyses. The Lenalidomide Information Sheet will be given to each patient receiving lenalidomide study therapy. The patient must read this document prior to starting lenalidomide study treatment and each time they receive a new supply of study drug.
* Social security cover
* Conditions of global RPP have to be fulfilled by all the patients
* The Lenalidomide Education and Counseling Guidance Document must be completed and signed by either a trained counselor or the Investigator at the participating clinical center prior to each dispensing of lenalidomide study treatment. A copy of this document must be maintained in the patient records.

Exclusion Criteria:

* Central nervous system involvement (cerebral CT scan is performed at the inclusion)
* One or more of the biological abnormalities :

Neutrophil count < 1,500/mm3 ; Platelet count < 60,000/mm3 ; Transaminases > 5 x upper limit of normal ; Total bilirubin > 2.0 mg/dl (34 µmol/L)/ conjugated bilirubin>0.8 mg/dL, except of haemolytic anemia ; Creatinine clearance < 50 mL /min ( measured or calculated according to the method of Cockcroft-Gault)

* Pregnant or lactating females, potentially childbearing females defined by sexually mature female who: 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months.
* Patients should not receive steroids continuously except for prednisone for tumoral flare treatment
* Uncontrolled infectious and thromboembolic diseases
* Subjects not willing to take deep venous thrombosis prophylaxis
* Prior history of malignancies unless the subject has been free of the disease for ≥5 years. Exceptions include basal cell skin carcinoma, carcinoma in situ of the cervix or of the breast
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Known seropositive for or active viral infection with HIV, Hepatitis B and C virus.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring parenteral antibiotics, uncontrolled diabetes mellitus as defined by the investigator
* Chronic symptomatic congestive heart failure (III or IV of the NYHA Classification for Heart Disease)
* Unstable angina pectoris, angioplasty or myocardial infarctions within 6 months
* Clinically significant cardiac arrhythmia that is symptomatic or requires treatment, or asymptomatic sustained ventricular tachycardia.
* Prior ≥ Grade 3 allergic reaction/hypersensitivity or desquamative rash while taking thalidomide
* Any standard or experimental anti-cancer drug therapy or radiation within 3 weeks of the initiation of study drug therapy.
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete response CR and partial response PR) at 6 months | 6 months after study treatment start
  Response will be assessed according to clinical and isotopic criteria.

SECONDARY OUTCOMES:
Overall response rate (complete response CR and partial response PR) at 12 months | 12 months after study treatment start
  Response will be assessed according to clinical and isotopic criteria.
Duration of response | Every 6 months
  Time between the first PR and progression
Progression-free survival | Every 6 months
  Time between the beginning of the treatment by lenalidomide and progression or death
Overall survival and disease specific survival | Evrey 6 months
Safety : description of adverse events occured including grade based on CTCAE v4.0 | Monthly during treatment duration (up to 12 months)
Quality of life | Every 2 months during treatment duration (up to 12 month)

CONTACTS AND LOCATIONS:
Overall Officials: Marie BEYLOT-BARRY, MD-PhD, Principal Investigator — University Hospital, Bordeaux; Eric FRISON, MD, Study Chair — Unité de Soutien Méthodologique à la Recherche clinique et épidémiologique; University Hospital, Bordeaux
Locations (24):
- France (24):
  - CHU Amiens, Hôpital Sud, Amiens
  - CHU Besançon, Hôpital Saint-Jacques, Besançon
  - AP-HP Hôpital Avicenne, Bobigny
  - AP-HP Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU de Clermont-Ferrand, Estaing, Clermont-Ferrand
  - AP-HP Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Le Bocage, Dijon
  - CHU de Grenoble, Grenoble
  - CHU de Lille Hôpital Claude Huriez, Lille
  - Centre Léon Bérard, Lyon
  - AP-HM Hôpital Nord, Marseille
  - CHRU de Montpellier Hôpital Saint-Eloi, Montpellier
  - CHU de Nantes, Hôtel Dieu, Nantes
  - CHU de Nice Groupe hospitalier l'Archet, Nice
  - AP-HP- Hôpital Saint Louis, Paris
  - AP-HP Groupe hospitalier Cochin, Paris
  - AP-HP Groupe hospitalier Bichat - Claude Bernard, Paris
  - AP-HP Hôpital Tenon, Paris
  - CHU de Bordeaux Hôpital du Haut Lévèque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Reims, Hôpital Robert Debré, Reims
  - CHU de Rouen, Hôpital Charles Nicolle, Rouen
  - CHU de Toulouse Hôpital Larrey, Toulouse
  - CHU de Tours- Hôpital Trousseau, Tours